CLINICAL TRIAL: NCT00876161
Title: Phase 1 Clinical Study With DAS181: Double-Blind, Randomized, Placebo-Controlled, Single Dose Escalation Study in Healthy Adults
Brief Title: DAS181 Single Dose Escalation Study in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ansun Biopharma, Inc. (Industry)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Patricia A. Meier, MD, Quintiles Phase One Services
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DAS181-1-02; Contract: HHSN266200600015CIb
Record Dates: First submitted 2009-04-03; First posted 2009-04-06 (Estimated); Last update posted 2019-08-02 (Actual); Status verified 2019-08

CONDITIONS: Healthy
Keywords: Healthy Adults
MeSH Terms: interventions — oplunofusp; Lactose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DAS181 (Experimental)
  Interventions: Drug: DAS181
- Lactose (Placebo Comparator)
  Interventions: Drug: Lactose

INTERVENTIONS:
Drug: DAS181 — DAS181 is formulated as dry powder and packaged in capsules containing DAS181. The delivered dose of DAS181 dry powder at each fill size is 5 mg, 10 mg and 20 mg.
  Arms: DAS181
Drug: Lactose
  Arms: Lactose

SUMMARY:
This study will evaluate the safety, tolerability, and systemic exposure of an experimental influenza (flu) treatment medication called DAS181. DAS181 is a dry powder that is administered via oral inhalation using a special device. Study participants will include healthy non-smoking males and females, ages 18-65. They will be given either DAS181 or placebo. Participants will remain in the clinic overnight to be watched for health changes for 24 hours after receiving the medication. Study procedures include: physical exams, chest x-rays, ECGs, lung function tests, collection of blood and urine samples, and throat swabs. Follow-up visits will occur on study days 2, 7, 14 and 30.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects in generally good health in the opinion of the investigator as determined by vital signs, medical history, and a targeted physical exam based on medical history.
* Subjects must be able to verbalize understanding of the consent form, provide written informed consent and verbalize willingness to complete study procedures
* Be 18 to 65 years of age (inclusive), in the past 12 months.
* Subjects must weigh at least 50 kg and must have a Body Mass Index (BMI) of no greater than 35.
* No recent history of smoking in the past two years regardless of clinical relevance.
* No history of alcoholism or alcohol abuse regardless of clinical relevance.
* Electrocardiogram (ECG) with no clinically significant abnormalities recorded at screening visit: PR interval within 120 and 200 ms, QRS interval < 120 ms, and QTc interval ≤ 440 ms.
* Blood pressure within normal limits (systolic 90-140mmHg; diastolic 50-90 mmHg) and heart rate between 45 and 100 beats per minute.
* Chest X-ray and FEV1 results show no clinically significant abnormalities.
* Negative HIV, HBV, and HCV screening tests.
* Hemoglobin within provided range (see Appendix 2).
* White blood cell count and platelet count within provided range (see Appendix 2).
* Alkaline phosphatase (ALKP), total bilirubin, alanine aminotransferase (ALT), aspartate aminotransferase (AST), creatinine phosphokinase (CPK), within provided range (see Appendix 2).
* Serum glucose within provided range (see Appendix 2). If non-fasting glucose is abnormal, a fasting glucose measurement may be measured in its place. If this is within the provided range, then subject may be enrolled.
* Serum creatinine within provided range (see Appendix 2).
* Activated partial thromboplastin time (APTT), Fibrinogen within provided range (see Appendix 2).
* Urine glucose, protein, and hemoglobin tested by dipstick urinalysis are negative or not greater than trace. Menstruating females failing inclusion due to positive urine dipstick hemoglobin may be retested following cessation of menses.
* Female subjects must be post-menopausal (one year or greater without menses), surgically incapable of childbearing, or practicing an acceptable method of birth control. Acceptable methods may include intrauterine device, spermicide and barrier, abstinence and hormonal contraception. A female subject must agree to practice an acceptable method of birth control during study period and for 12 weeks after study terminates. She must have had a negative serum pregnancy test during the screening visit and a negative urine pregnancy test on the day of treatment prior to study drug dosing.
* If male, agrees to use medically accepted form of contraception from time of enrollment to 12 weeks after study termination
* Subjects must test negative for drugs and alcohol

Exclusion Criteria:

* Have received any investigational drug or vaccine within 8 weeks prior to study drug dosing or have had a serious adverse reaction or hypersensitivity to any drug
* Have received blood products within 6 months of study enrollment
* Have been on a liquid protein diet in the last month.
* Are allergic or intolerant to lactose.
* Have sickle cell disease
* Have used prescription drugs, excluding hormonal contraception, within 7 days prior to admission (at the investigator's discretion) or non-prescription drugs (including herbal supplements) within 7 days prior to admission (at the investigator's discretion).
* Existence of any surgical, medical,or laboratory condition that, in the judgment of the clinical investigator, might interfere with the safety, distribution, metabolism or excretion of the drug
* Subjects with concurrent respiratory diseases (e.g., asthma, allergic rhinitis, chronic obstructive pulmonary disease, cystic fibrosis, or emphysema, anaphylaxis).
* Subjects who have experienced a previous episode of acute upper respiratory tract infection, pneumonia, otitis, bronchitis, or sinusitis within 2 weeks prior to screening.
* Subjects with concurrent sustained respiratory symptoms (running nose, sore throat, sneezing, coughing, or wheezing).
* Subjects who have an oral temperature above 37.8°C (100°F).
* Subjects with previous or current history of the following conditions: renal, hepatic, cardiac, pulmonary, hematologic, muscular, neurological, metabolic, or immunological disorders, hepatitis or cirrhosis, transplant recipients, HIV-infection, or other immunosuppressive illness.
* Subjects with cancer or history of hematologic malignancy. Cancer is defined as any active neoplastic diseases excluding noninvasive basal cell carcinoma.
* Subjects who have surgery within 30 days of initiation of the study.
* Female subjects who are pregnant or breast-feeding.
* Subjects who have donated or lost more than 500 mL of blood in the three months prior to screening.
* Subjects who have clinically significant medical or psychological conditions that would compromise the subject's safety, influence the results of the study, affect the subject's ability to participate in the study, or impair the subject's ability to provide informed consent.
* Subjects who have a history of drug dependence, or psychiatric illness within 2 years of study enrollment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2009-05-18 (Actual); Primary Completion 2009-12 (Actual); Study Completion 2010-05-23 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety, tolerability and pharmacokinetics of DAS181 dry powder inhalant single-dose treatment in healthy adults. | September 2009

CONTACTS AND LOCATIONS:
Locations (1):
- Quintiles Phase One Services, Overland Park, Kansas, United States

REFERENCES:
- See also: NexBio Inc — http://nexbio.com